CLINICAL TRIAL: NCT00152412
Title: A 4 Week Open, Multi-center Study Evaluating the Safety of Levocetirizine 1.25 mg b.i.d. Given as 0.5 mg/mL Oral Solution in 2 to 6 Year-old Children Suffering From Allergic Rhinitis.
Brief Title: Open Study to Evaluate the Safety of Levocetirizine in Young Children (2 - 6 Years) Suffering From Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A00385
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2009-09

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis, safety, levocetirizine, children; Xyzal
MeSH Terms: conditions — Rhinitis, Allergic | interventions — levocetirizine

INTERVENTIONS:
Drug: Levocetirizine oral solution

SUMMARY:
4 week open study to evaluate the safety of levocetirizine in young children (2 - 6 years) suffering from allergic rhinitis. As secondary objective, this study will assess the efficacy of the treatment by means of the T4SS (Total 4 symptoms scores of allergic rhinitis) and each of the 4 individual rhinitis symptom scores

ELIGIBILITY:
Inclusion Criteria:

* At Visit 1:

  * Male or female outpatients aged 2 to 6 years old.
  * Subjects suffering from allergic rhinitis (perennial and/or seasonal) and symptomatic as attested by the Daily Record Card (DRC).
* At Visit 2:

  * Respected wash-out periods for the forbidden medication.

Exclusion Criteria:

* • Presence of asthma requiring treatment by inhaled corticosteroids.

  * Atopic dermatitis or urticaria requiring antihistamine treatment or the administration of oral or topical corticosteroids, or any other disease requiring the administration of oral or topical corticosteroids, immunomodulatory drugs, anti-inflammatory, or cytotoxic drugs.
  * Use during the course of the study, or during the specific wash-out periods, of any of the following medications: intranasal or systemic corticosteroids (within 7 days), ketotifen (within 7 days), nedocromil or cromoglicate (within 7 days), loratadine and desloratadine (within 7 days), other antihistamines (within 3 days) or decongestants (per os, nasal spray, or drops - within 3 days), or any other concomitant medications that, in the opinion of the Investigator, interfered with the study.
  * Initiation or change of dose of an immunotherapy regimen during the course of the study.

Ages: 2 Years to 6 Years | Sex: All
Age Groups: Child
Enrollment: 30
Dates: Start 2004-06; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
To assess safety of levocetirizine 1.25 mg bid given as 0.5 mg/mL oral solution in 2 to 6 years old children suffering from allergic rhinitis over 4 weeks of treatment

SECONDARY OUTCOMES:
To assess efficacy of 1.25 mg levocetirizine 0.5 mg/mL oral solution bid in 2 to 6 years old children suffering from allergic rhinitis over 4 weeks by means of the T4SS and each of the 4 individual rhinitis
To describe the serum concentration of levocetirizine after 1,3 and 6 hours following the last treatment intake

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma